CLINICAL TRIAL: NCT04766398
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Phosphate Binder-combination, Parallel-group Comparative Study of KHK7791 in Hyperphosphatemia Patients on Hemodialysis
Brief Title: Phosphate Binder-combination Study of KHK7791 in Hyperphosphatemia Patients on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7791-005
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Hyperphosphatemia
Keywords: Tenapanor; Hyperphosphatemia; Hemodialysis
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHK7791 (Active Comparator): During the dosing period, subjects administer the study drug (KHK7791 or placebo) twice daily just before meals in a double blind. The starting dose of the study drug is 5 mg at a time, and the dose is adjusted in the range of 5, 10, 20, and 30 mg at a time based on the dose adjustment criteria described in the study protocol. Dosage adjustment is performed step by step.
  Interventions: Drug: KHK7791
- Placebo (Placebo Comparator): During the dosing period, subjects administer the study drug (KHK7791 or placebo) twice daily just before meals in a double blind. The starting dose of the study drug is 5 mg at a time, and the dose is adjusted in the range of 5, 10, 20, and 30 mg at a time based on the dose adjustment criteria described in the study protocol. Dosage adjustment is performed step by step.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK7791 — oral administration
  Arms: KHK7791
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of KHK7791 in combination with phosphate binders by comparing changes in serum phosphorus levels between hemodialysis patients with hyperphosphatemia receiving repeated administration of KHK7791 30 mg in combination with phosphate binders for 6 weeks and those receiving placebo in combination with phosphate binders.

ELIGIBILITY:
Inclusion Criteria:

1. Has voluntarily provided written informed consent to participate in the study.
2. Aged ≥ 20 years (expressed in completed years) at the time of providing informed consent.
3. Stable chronic renal failure patients who have undergone hemodialysis 3 times per week for at least 12 weeks until screening examination.
4. Dialysis conditions, excluding dry weight, should have been unchanged during the last 2 weeks before screening examination.
5. The prescribed drug and dosage regimen should have been unchanged during the last 4 weeks before screening examination.
6. Serum phosphorus levels should be in the range of ≥ 3.5 and ≤ 6.0 mg/dL at screening examination.
7. If on any vitamin D, calcimimetics regimen, bisphosphonate,calcitonin preparations, selective estrogen receptor modulators or teriparatide preparations then the prescribed drug and dosage regimen should have been unchanged for the last 4 weeks before screening examination.
8. Kt/V urea ≥ 1.2 at the most recent test in routine medical practice before screening examination.

Exclusion Criteria:

1. Peritoneal dialysis was performed within 12 weeks before screening examination.
2. iPTH >600 pg/mL (should be based on the most recent value from the patients' medical records, etc. before pre-enrollment)
3. Having concurrent or a history of inflammatory bowel disease (IBD) or diarrhea-predominant irritable bowel syndrome
4. History of gastrectomy or enterectomy or having undergone gastrointestinal tract surgery within 3 months before screening examination.
5. Subjects who used anti RANKL preparations within 6 weeks before screening examination.
6. Subjects who used anti-sclerostin antibody preparations within 12 weeks before screening examination.
7. Having concurrent severe heart disease or hepatic impairment.
8. Developed cerebrovascular disease requiring hospitalization within 6 months before screening examination.
9. Uncontrollable hypertension or diabetes.
10. Scheduled for living donor kidney transplant, change in the mode of dialysis, home hemodialysis, or change in the dialysis center (relocate to another hospital/clinic) during the study period.
11. Any diagnosis of and treatment of malignancy within 5 years before screening examination (excluding basal cell carcinoma or surgically resected intraepithelial carcinoma of uterine cervix).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Changes in serum phosphorous levels from baseline values at 8 weeks after the start of administration. | Week 8

SECONDARY OUTCOMES:
Changes in serum phosphorous levels from baseline values at each time point. | Dose period, Week 1, 2, 3, 4, 5, 6, 7, 8.
Achievement/failure of the target serum phosphorus level (serum phosphorus level: ≤ 6.0). | Dose period, Week 1, 2, 3, 4, 5, 6, 7, 8.
Time when the target serum phosphorus level (serum phosphorus level: ≤ 6.0) was achieved. | Dose period, Week 1, 2, 3, 4, 5, 6, 7, 8.
Achievement/failure of the target serum phosphorus level (serum phosphorus level: ≤ 5.5). | Dose period, Week 1, 2, 3, 4, 5, 6, 7, 8.
Time when the target serum phosphorus level (serum phosphorus level: ≤ 5.5) was achieved. | Dose period, Week 1, 2, 3, 4, 5, 6, 7, 8.
Concentrations of such as Ca × P product levels at each time point. | Dose period, Week 1, 2, 3, 4, 5, 6, 7, 8.
Changes of such as Ca × P product levels from baseline values at each time point. | Dose period, Week 1, 2, 3, 4, 5, 6, 7, 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Inoue Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No